CLINICAL TRIAL: NCT00756392
Title: MR Spectroscopy in Localized Prostate Cancer
Brief Title: Magnetic Resonance (MR) Spectroscopy in Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: GU-24315
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: 3T MR Spectroscopy; Prostate Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Procedure: 3T MR Spectroscopy

INTERVENTIONS:
Procedure: 3T MR Spectroscopy — A Magnetic Resonance Spectroscopy (MRS)study of a patient's prostate will be conducted with the 3 Tesla Philips Intera Nuclear Magnetic Resonance (NMR) scanner before and after filling the rectum with barium. Scan duration from Preparation to Completion will be approximately 30 minutes. The spectra will be acquired without and with the presence of Barium solution to compare to see if the latter is advantageous.

SUMMARY:
This study is designed to investigate whether filling the rectum with high density barium prior to a magnetic resonance spectroscopy (MRS)exam of the prostate improves the quality of the acquired spectrum. It is expected that the dense substance should help prevent air from entering the rectum and thus susceptibility artifacts in the obtained MRS data should be reduced. Ten patients with localized prostate cancer will be recruited for this study. There will be no change in treatment planning based on MRS study. Patient will receive standard radiation treatment prescribed by radiation oncologist.

DETAILED DESCRIPTION:
This study is designed to investigate whether filling the rectum with high density barium prior to a magnetic resonance spectroscopy (MRS) exam of the prostate improves the quality of the acquired spectrum. It is expected that the dense substance should help prevent air from entering the rectum and thus susceptibility artifacts in the obtained MRS data should be reduced. Ten patients with localized prostate cancer will be recruited for this study. There will be no change in treatment planning based on MRS study. Patient will receive standard radiation treatment prescribed by radiation oncologist.

An MRS study of each patient's prostate will be conducted with the 3 Tesla Philips Intera NMR (Nuclear Magnetic Resonance) scanners before and after filling the rectum with barium. Patients will be requested to take a mild laxative of their choice the night before the exam, and not to eat for 2-4 hours prior to the scan. To facilitate this, that patient's exam will be booked prior to lunch. Prior to the exam, the patient will be asked to empty their bladder and 40 mg of Buscopan will be administered to the patient (i.m. of i.v.) to reduce peristalsis, the presence of which degrades the quality of NMR scans. The patient will lie on a board designed to fit on the MR scanner patient bed and that holds one of the elements of the dual element phased array radiofrequency (RF) coil in place. The patient will be positioned such that the prostate is within the coil's field of view (preferably along its central axis); that is, the patient will lie on one element of the coil and the other element will be placed on top of the patients abdomen. An abdominal restraint will be placed around the patients abdomen to reduce breathing effects. After the patient has been centered in the magnet, MRI (Magnetic Resonance Imaging) images will be acquired to identify the tumor location. The positioning of the MRS voxel with the prostate will be carefully determined with the aid of a radiation oncologist. Preparation scans for the spectroscopy acquisition will be carried out prior to applying a PRESS (Point RESolved Spectroscopy) sequence that will be employed to obtain a proton (1H) spectrum of the prostate. The entire scan duration from preparation till completion will be approximately 30 minutes (5 minutes for patient positioning, 10 minutes for imaging and voxel placement, 5 minutes for spectroscope sequence preparation scans, and 10 minutes for spectrum acquisition). Following scan completion, the patient will have about 150 mL of Barium solution administered to the rectum. After standing for 3-4 minutes, the patient will like back on the NMR scanner bed and the same NMR procedure will be repeated again. The spectra acquired without and with the presence of Barium solution in the rectum will be compared to see if the latter situation is indeed advantageous.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Localized prostate cancer patients
* Signed informed consent form

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Imaging study to determine quality spectra on 3T MR | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Pervez, MD, FRCPC, Study Chair — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada